CLINICAL TRIAL: NCT00022152
Title: Phase II Trial of Oral Vinorelbine for the Treatment of Metastatic Breast Cancer in Patients >65 Years of Age: A Trial of Efficacy, Toxicity, and Patients' Perceived Preference for Oral Therapy
Brief Title: Vinorelbine in Treating Older Women With Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N003A; NCI-2012-02395 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000068790 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vinorelbine (Experimental): Patients receive oral vinorelbine once weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed at baseline and then after completion of the second course.
  Patients are followed every 3 months for 5 years.
  Interventions: Drug: vinorelbine tartrate

INTERVENTIONS:
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of vinorelbine in treating older women who have stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate in elderly women with stage IV breast cancer treated with oral vinorelbine.
* Determine the toxicity profile of this drug in these patients.
* Determine the time to progression in patients treated with this drug.
* Determine the quality of life of patients treated with this drug.
* Assess individual variation in responses (toxicity and/or activity), pharmacokinetic parameters, and/or biologic correlates due to genetic differences in enzymes involved in the transport, metabolism, and/or mechanism of action of this drug in these patients.

OUTLINE: Patients receive oral vinorelbine once weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then after completion of the second course.

Patients are followed every 3 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IV breast cancer
* Eligible to receive first- or second-line chemotherapy
* At least 1 unidimensionally measurable lesion

  * At least 20 mm in longest diameter
  * Must be completely outside prior irradiation port unless there is proof of progressive disease after completion of prior radiotherapy
* No untreated brain metastases

  * Current metastatic CNS disease allowed only if previously treated and clinically stable at study entry
* No meningeal carcinomatosis
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 65 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Total bilirubin no greater than 1.5 times upper limit of normal (ULN) OR
* Direct bilirubin normal if total bilirubin elevated or less than 2.5 times ULN because of Gilbert's syndrome

Renal:

* Creatinine no greater than 2 times ULN

Other:

* No grade 2 or greater peripheral neuropathy
* No other significant medical condition that would preclude study
* No active infection within the past 2 weeks
* No dysphagia or inability to swallow intact capsules

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No more than 1 prior chemotherapy regimen for metastatic disease
* No prior vinca alkaloids
* At least 4 weeks since other prior chemotherapy and recovered

Endocrine therapy:

* Prior hormonal therapy allowed
* No concurrent hormonal therapy

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to 25% or more of bone marrow
* At least 3 weeks since prior radiotherapy and recovered

Surgery:

* At least 3 weeks since prior major surgery

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-11; Primary Completion 2006-03 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
objective response rate | Up to 5 years

SECONDARY OUTCOMES:
time to progression | Up to 5 years
quality of life | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic
Locations (18):
- United States (18):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Baweja M, Suman VJ, Fitch TR, Mailliard JA, Bernath A, Rowland KM, Alberts SR, Kaur JS, Perez EA; NCCTG. Phase II trial of oral vinorelbine for the treatment of metastatic breast cancer in patients > or = 65 years of age: an NCCTG study. Ann Oncol. 2006 Apr;17(4):623-9. doi: 10.1093/annonc/mdj130. Epub 2006 Mar 6. PMID 16520332